CLINICAL TRIAL: NCT02807454
Title: A Phase 2, Multicenter, Open-label, Study to Determine the Safety and Efficacy for the Combination of Durvalumab (DURVA) and Daratumumab (DARA) (D2) in Subjects With Relapsed and Refractory Multiple Myeloma (RRMM)
Brief Title: A Study to Determine the Safety and Efficacy for the Combination of Durvalumab and Daratumumab in Relapsed and Refractory Multiple Myeloma
Acronym: FUSIONMM-003
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Health Authority request due to class effect
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDI4736-MM-003
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma
Keywords: Phase 2; Open-Label; Durvalumab; Daratumumab; Multiple Myeloma; Relapsed and Refractory (RRMM); FUSION MM-003; PD-L1
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — daratumumab; durvalumab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daratumumab Plus Durvalumab Treatment (Experimental): * Intravenous (IV) durvalumab at 1500mg on Day 1 or 2 of a 28-day cycle
  * IV daratumumab at 16mg/kg on days 1, 8, 15 and 22 at cycles 1-2; on days 1 and 15 at cycles 3-6; and on day 1 from cycle 7 onward
  Interventions: Drug: Daratumumab; Drug: Durvalumab
- Pomalidomide+ Daratumumab+ Durvalumab+ Dexamethasone Treatment (Experimental): * Intravenous (IV) durvalumab at 1500mg on Day 1 or 2 of a 28-day cycle
  * IV daratumumab at 16mg/kg on days 1, 8, 15 and 22 at cycles 1-2; on days 1 and 15 at cycles 3-6; and on day 1 from cycle 7 onward
  * oral POM at 4mg/day on days 1 to 21
  * oral/IV dex at 40mg/day (>75 years old) or 20mg/day (>75 years old) on days 1, 8, 15 and 22
  Interventions: Drug: Daratumumab; Drug: Durvalumab; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab
Drug: Durvalumab
Drug: Pomalidomide
  Arms: Pomalidomide+ Daratumumab+ Durvalumab+ Dexamethasone Treatment
Drug: Dexamethasone
  Arms: Pomalidomide+ Daratumumab+ Durvalumab+ Dexamethasone Treatment

SUMMARY:
This is an open-label, multicenter study to confirm the safety and efficacy of durvalumab + daratumumab (D2) in subjects with relapsed and refractory multiple myeloma. This study will also explore the safety and efficacy of the addition of pomalidomide + dexamethasone to durvalumab + daratumumab (PD3).

On 05 Sep 2017, a Partial Clinical Hold was placed on this study by the United States (US) Food and Drug Administration (FDA). The decision by the FDA was based on data related to risks of anti-programmed cell death-1 (PD-1) antibody, pembrolizumab, in combination with IMiDs® immunomodulatory drugs in patients with multiple myeloma. As a result, enrollment into this study has been discontinued. Subjects who are receiving clinical benefit, based on the discretion of the investigator, may remain on study treatment after being reconsented.

ELIGIBILITY:
Inclusion Criteria:

* Must have measurable disease as defined by m-protein or serum free light chain.
* Must have failed last line of treatment (refractory to last line of treatment).
* Must have achieved at least a minimal response (MR) to at least 1 prior anti-myeloma regimen before developing PD (relapsed)
* Has performance status of 0, 1, or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Must be at least 18 years of age

Exclusion Criteria:

* Has non-secretory multiple myeloma
* Has had prior anti-myeloma therapy within 2 weeks prior to study Day 1
* Has received prior therapy with an anti-programmed cell death 1 receptor (anti-PD-1), antiprogrammed death-ligand 1 (anti-PD-L1), anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways).
* Has received prior treatment with daratumumab or other anti-CD38 therapies previously
* Has undergone prior organ or allogeneic hematopoetic stem cell transplantation
* Has received autologous stem cell transplantation (ASCT) within 12 weeks before the date of randomization.
* Has received prior treatment with a monoclonal antibody within 5 half-lives of Study Day 1
* Has received investigational agents within 28 days or 5 half-lives (whichever is longer) of Study Day 1
* Has received live, attenuated vaccine within 30 days prior to Study Day 1
* Has chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) 50% of predicted normal
* Has moderate or severe persistent asthma within the past 2 years or uncontrolled asthma of any classification.
* Is positive for human immunodeficiency virus (HIV), chronic or active hepatitis B or active hepatitis A or C
* Has a prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥ 5 years (with the exception Basal cell carcinoma of the skin, Squamous cell carcinoma of the skin, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histologic finding of prostate cancer [T1a or T1b] or prostate cancer that is curative)
* Has clinical evidence of central nervous system (CNS) or pulmonary leukostasis, disseminated intravascular coagulation, or CNS multiple myeloma
* Has clinically significant cardiac disease
* Is a female who is pregnant, nursing, or breastfeeding, or who intends to become pregnant during the participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (64):
- United States (15):
  - City of Hope National Medical Center, Duarte, California
  - UCLA Division of Hematology Oncology, Los Angeles, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Local Institution - 007, Denver, Colorado
  - Emory University Hospital, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Center For Cancer and Blood Disorders, Bethesda, Maryland
  - Dana-Farber Partners Cancer Care, Inc., Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology Nashville Drug Development Unit, Nashville, Tennessee
  - Swedish Medical Center, Seattle, Washington
- Belgium (3):
  - AZ St-Jan Brugge Oostende AV, Bruges
  - Universitaire Ziekenhuizen Leuven Univeristy Hospitals Leuven, Leuven
  - Cliniques Universitaires UCL de Mont-Godine, Yvoir
- Canada (7):
  - Local Institution - 103, Saint John, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Local Institution - 104, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Local Institution - 101, Montreal, Quebec
  - MUHC Glen Site, Montreal, Quebec
- Denmark (6):
  - Local Institution - 552, Copenhagen
  - Rigshospitalet University Hospital, Copenhagen
  - Local Institution - 553, Odense
  - Odense University Hospital, Odense
  - Local Institution - 551, Vejle
  - Vejle Hospital, Vejle
- Germany (6):
  - Universitatsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Local Institution - 203, Heidelberg
  - Universitatsklinikum Heidelberg, Heidelberg
  - University Hospital Tubingen, Tübingen
  - Local Institution - 201, Würzburg
  - Universitatsklinikum Wuerzburg, Würzburg
- Italy (8):
  - Local Institution - 354, Bologna
  - Policlinico S. Orsola - Malpighi, Bologna
  - A.O.U. Maggiore della Carità, Novara
  - Local Institution - 353, Novara
  - Azienda Ospedaliera di Padova, Padua
  - Local Institution - 355, Padua
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello, Palermo
  - A.O. Universitaria Ospedale S.Chiara Dip.Oncologia, Div. Ematologia, Pisa
- Spain (7):
  - Hospital Durán i Reynals - Instituto Catalàn de Oncologìa ICO, Barcelona
  - Local Institution - 453, Barcelona
  - Hospital de Cabuenes, Gijón
  - Local Institution - 451, Gijón
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Local Institution - 452, Madrid
  - Hospital 12 de Octubre, Madrid
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Local Institution - 501, Lund
  - Skanes Universitetssjukhus Malmo, Lund
  - Local Institution - 502, Stockholm
  - Karolinska Universitetssjukhuset - Huddinge, Stockholm
- United Kingdom (7):
  - St. Bartholomew's and The Royal London Hospital, London
  - Christie Hospital, Manchester
  - Local Institution - 252, Oxford
  - Oxford University Hospitals NHS Trust- Churchill Hospital-Oxford Centre for Respiratory Medicine, Oxford
  - Local Institution - 253, Sutton (Surrey)
  - Royal Marsden Hospital, Sutton (Surrey)
  - The Royal Wolverhampton Hospital NHS Trust, Wolverhampton

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either Durvalumab + Daratumumab (D2) or Durvalumab + Daratumumab + Pomalidomide + Dexamethasone (PD3). 32 participants were treated in the Simon Stage 1: D2 arm. No participants enrolled in the Simon Stage 2: D2 arm. 5 participants treated in the PD3 arm.
Groups:
- Simon Stage 1: D2 Arm: Durvalumab 1500 mg + Daratumumab 16 mg/kg were administered intravenously within a 28-day cycle for a maximum of 60 cycles. POM + DEX could be added to the D2 regimen, at the investigator's discretion, upon confirmed progressive disease for participants who had at least 2 cycles of D2.
- PD3 Arm: Durvalumab 1500 mg IV + Daratumumab 16 mg/kg IV + Pomalidomide 4 mg/day Oral + Dexamethasone 40 mg Oral (20 mg for > 75 Years Old) administered within a 28-day cycle for a maximum of 22 cycles
Period: Overall Study
Arm/Group | Simon Stage 1: D2 Arm | PD3 Arm
Started | 32 | 5
Participants in the D2 Arm Who Also Received Pomalidomide + Dexamethasone | 7 | 0
Completed | 0 | 0
Not Completed | 32 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Progressive Disease | 30 | 3
Not completed — Other Reasons | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simon Stage 1: D2 Arm | PD3 Arm | Total
Number analyzed (Participants) | 32 | 5 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (7.58) | 63 (5.66) | 63.2 (7.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 1 | 14
  Male | 19 | 4 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 32 | 5 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 31 | 5 | 36
    Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Tumor response of partial response (PR) or better was assessed using the International Myeloma Working Group (IMWG) Uniform Response Criteria. ORR was calculated as the percent of responders (multiplied by 100). Partial response required ≥ 50% reduction of serum M-Protein and reduction in 24-hour urinary M protein by ≥ 90% or to < 200 mg per 24 hours.
Time Frame: From first dose to up to approximately 66 months
Population: All enrolled participants who received at least 1 dose of the study medication, and who have measurable disease at baseline and at least 1 postbaseline efficacy assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Simon Stage 1: D2 Arm | PD3 Arm
Number analyzed (Participants) | 32 | 4
Percentage of participants | 53.1 | 75.0

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants who experienced at least one adverse event. An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening (i.e., any clinically significant adverse change in the frequency or intensity of a preexisting condition should be considered an AE.
Time Frame: From first dose to 90 days after last dose (up to approximately 58 months)
Population: All participants who received at least 1 dose of the study medications.
Measure: Count of Participants; unit: Participants
Arm/Group | Simon Stage 1: D2 Arm | PD3 Arm
Number analyzed (Participants) | 32 | 5
Participants | 31 | 5

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of participants who experienced at least one serious adverse event. An SAE is any AE occurring at any dose that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, constitutes an important medical event.
Time Frame: From first dose to 90 days after last dose (up to approximately 58 months)
Population: All participants who received at least 1 dose of the study medications.
Measure: Count of Participants; unit: Participants
Arm/Group | Simon Stage 1: D2 Arm | PD3 Arm
Number analyzed (Participants) | 32 | 5
Participants | 17 | 2

4. Secondary Outcome: Time-To-Response (TTR)
Description: Time-to-response is calculated as the time from enrollment to the first date of documented response (partial response or better). Tumor response of partial response (PR) or better was assessed using the International Myeloma Working Group (IMWG) Uniform Response Criteria. Partial response required ≥ 50% reduction of serum M-Protein and reduction in 24-hour urinary M protein by ≥ 90% or to < 200 mg per 24 hours. For those participants where POM + DEX were added, time-to-response was calculated from the date POM and DEX were added to the first date of documented response (PR or better).
Time Frame: From enrollment to earliest documented response (up to approximately 66 months)
Population: All enrolled participants who received at least 1 dose of the study medication, and who have measurable disease at baseline and at least 1 postbaseline efficacy assessment in the D2, D2 + Pomalidomide + Dexamethasone, and PD3 arms.
Measure: Median (Full Range); unit: Weeks
Groups:
- Simon Stage 1: D2 Arm: Durvalumab 1500 mg + Daratumumab 16 mg/kg were administered intravenously within a 28-day cycle for a maximum of 60 cycles
- Simon Stage 1: D2 + Pomalidomide + Dexamethasone: Durvalumab 1500 mg IV + Daratumumab IV 16 mg/kg + Pomalidomide 4 mg/day Oral + Dexamethasone 40 mg Oral (20 mg for > 75 Years Old) were administered within a 28-day cycle for a maximum of 60 cycles
Arm/Group | Simon Stage 1: D2 Arm | Simon Stage 1: D2 + Pomalidomide + Dexamethasone | PD3 Arm
Number analyzed (Participants) | 32 | 7 | 4
Weeks | 4.29 [4.0 to 12.0] | 5.07 [4.1 to 8.1] | 8.14 [4.3 to 8.3]

5. Secondary Outcome: Kaplan-Meier Estimate of Duration of Response (DOR) - Simon Stage 1: D2 Arm
Description: Duration of response was calculated as the time from the earliest date of documented response (PR or better) to the earliest date of disease progression as determined by the investigator. For those participants where POM + DEX was added, duration of response was calculated as the time from the earliest date of documented response after POM + DEX was added (PR or better) to the earliest date of disease. Tumor response of partial response (PR) or better was assessed using the International Myeloma Working Group (IMWG) Uniform Response Criteria. Partial response required ≥ 50% reduction of serum M-Protein and reduction in 24-hour urinary M protein by ≥ 90% or to < 200 mg per 24 hours. Progressive Disease required increase of 25% from lowest response value in the serum M-component (absolute increase must be ≥ 0.5 g/dL) and/or urine M-component (absolute increase must be ≥ 200 mg/24 h).
Time Frame: From the earliest date of documented response (PR or better) to earliest date of progressive disease (up to approximately 66 months)
Population: All enrolled participants with a partial response or better, who received at least 1 dose of the study medication, and who have measurable disease at baseline and at least 1 postbaseline efficacy assessment. Pre-specified for data to be collected only in D2 and D2 + Pomalidomide + Dexamethasone arms.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Simon Stage 1: D2 + Pomalidomide + Dexamethasone: Durvalumab 1500 mg IV + Daratumumab 16 mg/kg IV + Pomalidomide 4 mg/day Oral + Dexamethasone 40 mg Oral (20 mg for > 75 Years Old) were administered within a 28-day cycle for a maximum of 60 cycles
Arm/Group | Simon Stage 1: D2 Arm | Simon Stage 1: D2 + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 32 | 7
Months | 8.31 [3.7 to 11.1] | 8.41 [3.7 to 12.0]

6. Secondary Outcome: Kaplan-Meier Estimate of Duration of Response (DOR) - PD3 Arm
Description: Duration of response was calculated as the time from the earliest date of documented response (PR or better) to the earliest date of disease progression as determined by the investigator. For those participants where POM + DEX was added, duration of response was calculated as the time from the earliest date of documented response after POM + DEX was added (PR or better) to the earliest date of disease progression as determined by the investigator. Participants who are alive or lost to follow-up will be censored on the last-known-to-be-alive date. Tumor response of partial response (PR) or better was assessed using the International Myeloma Working Group (IMWG) Uniform Response Criteria. Partial response required ≥ 50% reduction of serum M-Protein and reduction in 24-hour urinary M protein by ≥ 90% or to < 200 mg per 24 hours.
Time Frame: as for outcome 5
Population: All enrolled participants with a partial response or better, who received at least 1 dose of the study medication, and who have measurable disease at baseline and at least 1 postbaseline efficacy assessment. Pre-specified for data to be collected only in the PD3 arm.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | PD3 Arm
Number analyzed (Participants) | 4
Months | 7.62 [6.7 to 17.5]

7. Secondary Outcome: Kaplan-Meier Estimate of Progression-Free Survival (PFS) - Simon Stage 1: D2 Arm
Description: Progression-free survival was calculated as the time between the enrollment to the first documentation of progressive disease or death from any cause during study, whichever occurs earlier using the International Myeloma Working Group (IMWG) Uniform Response Criteria. Progressive Disease required increase of 25% from lowest response value in the serum M-component (absolute increase must be ≥ 0.5 g/dL) and/or urine M-component (absolute increase must be ≥ 200 mg/24 h).
Time Frame: From enrollment to first documentation of progressive disease or death from any cause during study, whichever occurs earlier (up to approximately 66 months)
Population: All participants who received at least 1 dose of the study medications. Pre-specified for data to be collected only in D2 and D2 + Pomalidomide + Dexamethasone arms.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Simon Stage 1: D2 Arm | Simon Stage 1: D2 + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 32 | 7
Months | 5.74 [2.0 to 6.5] | 8.05 [3.7 to 12.9]

8. Secondary Outcome: Kaplan-Meier Estimate of Progression-Free Survival (PFS) - PD3 Arm
Description: as for outcome 7
Time Frame: as for outcome 7
Population: All participants who received at least 1 dose of the study medications. Pre-specified for data to be collected only in the PD3 arm.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | PD3 Arm
Number analyzed (Participants) | 5
Months | 9.02 [6.9 to 18.5]

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) - Simon Stage 1: D2 Arm
Description: Pharmacokinetics of Durvalumab derived from serum concentration versus time data.
Time Frame: Cycle 1 - Days 2, 8, 15, 22
Population: All participants who received at least 1 dose of study medication and who have at least 1 measurable plasma concentration. Cmax was a pre-specified secondary outcome measure in the Simon Stage 1: D2 arm only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Simon Stage 1: D2 Arm
Number analyzed (Participants) | 30
ug/mL | 315.806 (34.832)

10. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) - Simon Stage 1: D2 Arm
Description: Pharmacokinetics of Durvalumab derived from serum concentration versus time data.
Time Frame: Cycle 1 - Days 2, 8, 15, 22
Population: All participants who received at least 1 dose of study medication and who have at least 1 measurable plasma concentration. Tmax was a pre-specified secondary outcome measure in the Simon Stage 1: D2 arm only.
Measure: Median (Full Range); unit: Hour
Arm/Group | Simon Stage 1: D2 Arm
Number analyzed (Participants) | 30
Hour | 1.150 [1.03 to 1.83]

11. Secondary Outcome: Area Under the Plasma Concentration-Time Curve to the Last Measurable Plasma Concentration [AUC(0-Last)] - Simon Stage 1: D2 Arm
Description: Pharmacokinetics of Durvalumab derived from serum concentration versus time data.
Time Frame: Cycle 1 - Days 2, 8, 15, 22
Population: All participants who received at least 1 dose of study medication and who have at least 1 measurable plasma concentration. [AUC(0-Last)] was a pre-specified secondary outcome measure in the Simon Stage 1: D2 arm only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*ug/mL
Arm/Group | Simon Stage 1: D2 Arm
Number analyzed (Participants) | 30
Hour*ug/mL | 77831.751 (48.535)

12. Secondary Outcome: Area Under the Plasma Concentration-Time Curve in 1 Dosing Interval [AUC(TAU)] - Simon Stage 1: D2 Arm
Description: Pharmacokinetics of Durvalumab derived from serum concentration versus time data.
Time Frame: Cycle 1 - Days 2, 8, 15, 22
Population: All participants who received at least 1 dose of study medication and who have at least 1 measurable plasma concentration. [AUC(TAU)] was a pre-specified secondary outcome measure in the Simon Stage 1: D2 arm only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*ug/mL
Arm/Group | Simon Stage 1: D2 Arm
Number analyzed (Participants) | 28
Hour*ug/mL | 83966.099 (46.115)

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from the participant's first dose to their study completion (up to approximately 66 months). SAEs and Other AEs were assessed from first dose to 90 days after last dose of study therapy (up to approximately 58 months).
Arm/Group | Simon Stage 1: D2 Arm | PD3 Arm
All-Cause Mortality (participants affected / at risk) | 11/32 | 4/5
Serious Adverse Events (participants affected / at risk) | 17/32 | 2/5
Other Adverse Events (participants affected / at risk) | 31/32 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simon Stage 1: D2 Arm (N=32) | PD3 Arm (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Cellulitis streptococcal (Infections and infestations) | 1 | 0
Corynebacterium infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simon Stage 1: D2 Arm (N=32) | PD3 Arm (N=5)
Anaemia (Blood and lymphatic system disorders) | 16 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 1
Lymphopenia (Blood and lymphatic system disorders) | 8 | 1
Neutropenia (Blood and lymphatic system disorders) | 15 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0
Cataract (Eye disorders) | 2 | 0
Conjunctival irritation (Eye disorders) | 0 | 1
Ophthalmic vein thrombosis (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 8 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1
Asthenia (General disorders) | 3 | 1
Chills (General disorders) | 2 | 1
Fatigue (General disorders) | 4 | 2
Gait disturbance (General disorders) | 0 | 1
Influenza like illness (General disorders) | 4 | 0
Mucosal inflammation (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Oedema (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 3 | 1
Pyrexia (General disorders) | 9 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Oral candidiasis (Infections and infestations) | 1 | 1
Pneumococcal infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 6 | 2
Sinusitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 8 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 0
International normalised ratio increased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 4 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 0
Sciatica (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 5 | 1
Restlessness (Psychiatric disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
This study stopped enrolling participants on 05-Sep-2017 and was terminated earlier than planned on 03-Jan-2022. This results disclosure report provides outputs from the Simon Stage 1: D2 and PD3 arms. Simon Stage 2: D2 did not enroll any participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT02807454/Prot_SAP_000.pdf